CLINICAL TRIAL: NCT00568399
Title: The Effect of Sodium Thiosulfate Treatment on Vascular Calcification in End Stage Renal Failure Patients
Brief Title: Sodium Thiosulfate Treatment of Vascular Calcification in ESRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRPO 07-0331
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Results first posted 2012-11-06 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Complication of Hemodialysis; Cardiovascular Diseases
Keywords: Coronary; Calcification; Dialysis; Thiosulfate; Cardiovascular
MeSH Terms: conditions — Cardiovascular Diseases; Calcinosis | interventions — sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active Treatment (Experimental): This is the only arm and involves active treatment with sodium thiosulfate in those subjects with high coronary artery calcium scores.
  Interventions: Drug: sodium thiosulfate

INTERVENTIONS:
Drug: sodium thiosulfate — sodium thiosulfate 12.5-25 gm/M2 after each thrice weekly hemodialysis treatments for 5 months.

SUMMARY:
Cardiovascular disease is the major cause of death in the hemodialysis population and calcification of the major arteries (coronary, aorta, and carotid) are a play a central role in this process. The major causes of the calcification are many, including high levels of phosphorus, low levels of inhibitors of calcification, positive calcium balance, and oxidative stress. Once vascular calcification is present, it is usually progressive. There is no known treatment to reverse established vascular calcification.

Sodium thiosulfate has been used extensively and safely to treat calcific uremic arteriopathy (a disease, in part due to calcification of small arteries) in dialysis patients. It increases the solubility of calcium by up to 100,000 fold and is also a potent anti-oxidant. It therefore has to potential to also decrease the amount of calcium in large arteries in dialysis patients and, hence improve survival.

We will study hemodialysis (HD) patients at high risk for cardiovascular disease and death by obtaining a multidetector computerized tomography (MDCT) Scan of the coronary arteries, carotid arteries and aorta and an assessment of coronary artery stenoses by a simultaneous intravenous infusion of contrast. At the same setting, we will perform tests of pulse wave velocity (PWV) and carotid ultrasound carotid intima-media thickness(CIMT)studies. In those patients at high risk for cardiovascular death, defined as a coronary artery calcification score (CACS)of greater than 50, sodium thiosulfate at a dose of 12.5-25 gm/1.73 M2 will be infused over 15-30 minutes after each dialysis treatment for 5 months. The above studies will then be repeated.

DETAILED DESCRIPTION:
Hypothesis 1: The treatment of HD patients with high CAC scores with sodium thiosulfate for 5 months will decrease the amount of calcium in their coronary arteries.

Patients who are at high risk for having coronary calcification (history of MI, ischemic heart disease, peripheral or carotid artery disease) will be selected to undergo testing. We will recruit 60 HD patients receiving treatment in our units to undergo MDCT scanning along with non-invasive testing of PWV and CIMT. Assuming that 60% will have a CAC score of ≥50, 36 patients will be treated with sodium thiosulfate. We will administer 25% sodium thiosulfate solution (American Reagent Laboratories, Shirley, NY) at a dose of 12.5-25g/1.73m2 per over 15-30 minutes after each hemodialysis session for a total of 60 treatments (5 months). Assuming a 35% attrition rate, 23 patients will complete the entire protocol and undergo a repeat study of the initial battery of tests.

Rationale for treatment with sodium thiosulfate: Sodium thiosulfate, used as an antidote for cyanide poisoning for more than a century, is also an anti-oxidant, and binds with calcium to form a highly soluble calcium thiosulfate salt. The solubility of calcium thiosulfate salt is 250-100,000 fold higher than calcium oxalate or calcium phosphate salt. It has been used to treat recurrent calcium kidney stones and tumoral calcinosis (ectopic calcification usually around joints). It has also been used successfully in treating calcific uremic arteriopathy, a disease of small artery and soft tissue calcification, in several studies of dialysis patients and in our own experience of 5 patients. By 2 months there is radiological evidence of reduction in soft tissue calcification. Unpublished data also have demonstrated regression of established aortic calcification in uremic rats.

Sodium thiosulfate is a FDA approved medication for the treatment of cyanide poisoning. It is classified by the FDA as "generally recognized as safe". There are no known contraindications. The only side effects reported during intravenous (IV) administration in ESRD patients are nausea, vomiting and hyperosmia during the administration, which can be alleviated by pre-administration of anti-emetic medications. Sodium thiosulfate is slowly given through the dialysis venous line toward the end of HD treatments. The selected dose for this pilot study is the same as that used for the treatment of calcific uremic arteriopathy.

We will freeze 10 ml of serum obtained prior to and then monthly during treatment for subsequent analyses. Included in the analysis will be Fetuin-A levels but other relevant markers will be considered. Blood will also be frozen for future genomic studies.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patient with thrice weekly treatments
* Coronary artery calcium score greater than 50
* Age greater than 18
* Compliant with hemodialysis treatments
* Informed consent

Exclusion Criteria:

* Allergy to sodium thiosulfate
* Pregnancy
* Incarceration
* Enrollment in another study
* Life expectancy less than 5 months
* Expectation of recovery of renal function
* Urine output of greater than 200 ml/day or contrast allergy will not receive intravenous contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Delmez, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients treated with chronic hemodialysis for ESRD at 2 Washington University units were recruited to undergo a battery of cardiovascular tests including CT quantitation (MDCT) of vascular calcification and possible treatment with sodium thiosulfate (see Am J Nephrol 2011;33:131-138)
Pre-assignment Details: All patients with a coronary artery calcium score of greater than 50 Angstrom scores were begun on treatment with sodium thiosulfate after each dialysis for 5 months and the battery of cardiovascular tests were repeated in those who completed the 5 months of treatment.
Groups:
- Sodium Thiosulfate: Treatment with sodium thiosulfate after each dialysis for 5 months and the battery of cardiovascular tests were repeated in those who completed the 5 months of treatment.subjects with high coronary artery calcium scores.
Period: Overall Study
Arm/Group | Sodium Thiosulfate
Started | 37
Completed | 22 (Of 48 subject enrolled, 37 initiated sodium thiosulfate treatment. 22 completed the entire protocol)
Not Completed | 15
Not completed — Death | 2
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Thiosulfate
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Annualized Coronary Calcium Volume Score After Treatment With Sodium Thiosulfate.
Description: We will compare the annualized coronary calcium volume score obtained at the baseline CT of the coronary arteries with another CT obtained of the same coronary arteries following 5 months of sodium thiosulfate treatment.
Time Frame: 5 months
Population: This is a feasibility study and all eligible participants were invited to participate. Out of the 48 participates that started, but only 22 completed.
Measure: Geometric Mean (Standard Deviation); unit: mm3/year
Groups:
- Sodium Thiosulfate: Treatment with sodium thiosulfate after each dialysis for 5 months
Arm/Group | Sodium Thiosulfate
Number analyzed (Participants) | 22
mm3/year | 6.6 (9.7)
Statistical Analysis 1: Comparison: Sodium Thiosulfate; This was a pilot study without a control group. There were no power calculations (see manuscript); Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney) — Coronary calcium score after treatment compared to baseline; Mean Difference (Final Values) = 9.2, Standard Deviation 0.987

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Sodium Thiosulfate
Serious Adverse Events (participants affected / at risk) | 2/37
Other Adverse Events (participants affected / at risk) | 5/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Thiosulfate (N=37)
Death due to retroperitoneal bleed (Renal and urinary disorders) | 1 (1)
Death due to sepsis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Thiosulfate (N=37)
Nausea (Gastrointestinal disorders) | 5

LIMITATIONS AND CAVEATS:
This study did not enroll a prospective, randomized, placebo controlled, double-blind control group; therefore conclusive statements about the risks and benefits of thiosulfate cannot be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes